CLINICAL TRIAL: NCT03833999
Title: Mode of Action of Ondansetron, a 5-HT Receptor 3 Antagonist, in Lactulose Induced Diarrhoea
Acronym: MOLID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 85-1807
Record Dates: First submitted 2019-01-07; First posted 2019-02-07 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-02

CONDITIONS: Motility Disorder of Intestine; Ondansetron; Small Bowel Water
Keywords: ondansetron; small bowel water
MeSH Terms: interventions — Ondansetron; Lactulose

STUDY DESIGN:
Intervention Model Description: double-blind, two-period, two-treatment crossover trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron and lactulose (Experimental): Ondansetron 8mg three times daily for 48 hours lactulose 20ml twice daily for 48 hours Serial abdominal MRI imaging
  Interventions: Drug: Ondansetron 8mg; Diagnostic Test: abdominal MRI; Drug: Lactulose
- Placebo and lactulose (Placebo Comparator): placebo oral capsule, one three times daily for 48 hours lactulose 20ml twice daily for 48 hours Serial abdominal MRI imaging
  Interventions: Diagnostic Test: abdominal MRI; Drug: Lactulose; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ondansetron 8mg — ondansetron, a 5HT3 receptor antagonist used clinically in nausea and vomiting
  Arms: Ondansetron and lactulose
Diagnostic Test: abdominal MRI — serial MRIs on day 1 and day 3 of the study, at baseline and 2 hours apart 0-6 hours after meal ingestion on day 1 and 0-4 hours after the meal on day 3
Drug: Lactulose — Participants will receive 20mls lactulose twice daily for 48 hours prior to the third study day
Drug: Placebo oral capsule — overcoated placebo tablet, identical to the ondansetron
  Arms: Placebo and lactulose

SUMMARY:
This is a double-blind, two period, two treatment crossover trial of ondansetron verses placebo studying the effects of ondansetron in the small and large bowel, specifically its effects on the amount of water in the gut, measured by MRI.

DETAILED DESCRIPTION:
If participants interested to take part the investigators will ask some questions to check participants are eligible to take part. Part of this involves measuring height, weight and having an electrocardiogram (ECG) to assess the heart. This is non-invasive and is achieved by attaching stickers across participants' chest. If participants are eligible the investigators will invite them to join the study, asked to sign a consent form and arrange for them to come to 4 study days.

Study Days The study days take place at the 3T Acheiva MRI scanner at the Sir Peter Mansfield Imaging Centre. This is located on the University Park campus.

The day before each scanning day participants will be asked to eat and drink as normal, avoiding beans or pulses and abstain from alcohol. The investigators ask that participants avoid strenuous exercise, and if they smoke to continue as normal.

On the morning of the day 1 of the study participants should come to the MRI scanner around 8 o'clock in the morning. They should not have anything to eat or drink at all, unless they need a sip of water to swallow essential medicines. The investigators will confirm that it is still safe for participants to be scanned and participants will then change into surgical scrubs (provided) to begin the study.

Participants will be randomly assigned to take either ondansetron, the anti-sickness tablet, for the first 2 visits or a dummy tablet (placebo) three times daily. They will be overcoated tablets so that neither participants nor the research team can tell which one it is.

Participants will then have an MRI scan, during which the investigators will scan the body in different ways. A separate information sheet tells participants more about this.

After these are done the investigators will give participants a meal supplement drink called Fortisip. Participants will have around 10 minutes to finish the drink. As soon as participants finish the MRI will be repeated. Participants will then have 3 further MRI scans, 2, 4 and 6 hours after the meal. After the last scan the investigators will give participants another dose of either the ondansetron or the placebo, and 20mls of a laxative called lactulose. The investigators will provide participants with tablets and the laxative for the following day at home.

Day 2 of the study participants can have a normal day at home, however the investigators ask that participants refrain from strenuous exercise, avoid alcohol, beans and pulses and continue a usual smoking habit if applicable. Participants are asked to take the tablet (either ondansetron or placebo) three times a day (in the morning, midday and evening) and 20mls of the laxative in the morning and evening. They are also asked to take 5 MRI marker tablets at 8pm, and take a timestamped photo or video so the investigators can ensure these are taken at the correct time. The marker tablets will be used to measure the speed of food along the gut on the scan on day 3.

On day 3 participants are asked to return for another day of scanning at the Sir Peter Mansfield Imagine Centre. Again, participants should come to the MRI scanner around 8 o'clock in the morning. They should not have anything to eat or drink at all, unless a sip of water is needed to swallow essential medicines. The investigators will re-confirm that it is still safe for participants to be scanned and participants will then change into surgical scrubs (provided) to begin the study.

Participants will receive a further dose of the ondansetron or placebo tablet, then have an MRI scan before drinking the same Fortisip meal supplement and the lactulose. Once participants have finished the drink they will have 2 further MRI scans, 2 and 4 hours after the meal. Participants can then leave for the day.

The investigators ask that participants come back to repeat the above 3 day procedure once more, taking the alternative tablet the second time around. Study periods will normally be one week apart. It is very important that participants attend both study periods as the investigators will compare the results from one week to the other.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* able to give informed consent

Exclusion Criteria:

* Pregnancy declared by candidate
* History declared by the candidate of pre-existing gastrointestinal disorder that may affect bowel function, congenital long QT syndrome or QTc >450msecs for males or 470 msecs for female on screening ECG.
* A positive diagnosis of irritable bowel syndrome based on the Rome IV criteria questionnaire
* Reported history of previous resection of the oesophagus, stomach or intestine (excluding appendix)
* Intestinal stoma
* Any medical condition making participation potentially compromising participation in the study e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner, known allergy to one of the food products
* Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* Will not agree to dietary restrictions required during the MRI study day
* Unable to stop drugs known to alter GI motility including mebeverine, opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants will be recorded but will not be an exclusion criteria)
* Inability to lie flat or exceed scanner limits of weight <120kg
* Poor understanding of English language
* Participation in night shift work the week prior to the study day. Night work is defined as working between midnight and 6.00 AM
* Participation in any medical trials for the past 3 months
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
small bowel water content | 0-6 hours post meal
  Change from baseline in area under the curve (AUC) small bowel water content

SECONDARY OUTCOMES:
small bowel motility (global motility score, arbitrary units) | 2 and 4 hours postprandially
  Change from baseline motility over the study using cine MRI. An increased value indicates increased small bowel motility
Weighted average position score (WAPS) | baseline on day 3
  MRI method of assessing colonic transit using MR marker pills ingested 12 hours before the scan. A lower value indicates faster whole gut transit
T1 of the ascending colon (T1AC) | baseline on day 3
  MRI measure of water content in the ascending colon.Change from baseline in AUC T1AC from 0-4 hours. A higher value indicates more watery ascending colon content.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans for sharing IPD